CLINICAL TRIAL: NCT01004055
Title: Efficacy of the PROCELLERA Wound Dressing in the Healing of Wounds After Curettage and Electrodesiccation of Skin Lesions
Brief Title: Efficacy Study of a Bioelectric Dressing to Treat Wounds Caused by Curettage and Electrodesiccation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vomaris Innovations (Industry)
Responsible Party: Scott Sheftel, MD, Sheftel Associates Dermatology, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XSMP-011
Record Dates: First submitted 2009-10-27; First posted 2009-10-29 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Wound Healing; Wound Infection
Keywords: Wound; Skin lesion; Antimicrobial; Bioelectric
MeSH Terms: conditions — Wound Infection; Wounds and Injuries | interventions — Acticoat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Procellera™ Wound Dressing (Experimental)
  Interventions: Device: Procellera™ Antimicrobial Wound Dressing
- ACTICOAT™ (Active Comparator)
  Interventions: Drug: ACTICOAT™ Antimicrobial Barrier Dressing
- Mepilex® Ag (Active Comparator)
  Interventions: Drug: Mepilex® Ag Silver Foam Dressing

INTERVENTIONS:
Device: Procellera™ Antimicrobial Wound Dressing — Dressing indicated for partial and full-thickness wounds. Dressing changes every 2-3 days, more frequently if needed
  Other Names: PROCELLERA™, PROSIT™, Bioelectric Wound Dressing
  Arms: Procellera™ Wound Dressing
Drug: ACTICOAT™ Antimicrobial Barrier Dressing — Dressing changes every 2-3 days, more frequently if needed
  Other Names: ACTICOAT™
  Arms: ACTICOAT™
Drug: Mepilex® Ag Silver Foam Dressing — Dressing changes every 2-3 days, more frequently if needed
  Other Names: Mepilex® Ag
  Arms: Mepilex® Ag

SUMMARY:
The purpose of this study is to determine whether a bioelectric wound dressing, a silver-coated dressing, or a silver-foam dressing are effective in the treatment of wounds resulting from curettage and electrodesiccation of skin lesions.

ELIGIBILITY:
Inclusion Criteria:

* If female, must either be not of childbearing potential or if they are of childbearing potential must have a negative urine pregnancy test
* Wound size greater than 1x1cm
* Wound must be ≥5 cm away from all other wounds
* Wound size must not be diminished in size greater than 10% between enrollment in study and the prescreening
* Participant agrees to participate in follow-up evaluation
* Participant must be able to read and understand informed consent, and sign the informed consent

Exclusion Criteria:

* Concurrent participation in another clinical trial that involves an investigational drug or device that would interfere with this study
* Participant is to receive another topical antimicrobial agent other than the study dressing
* Participant with sensitivity or adverse reactions to silver or zinc
* Pregnancy or nursing an infant or child
* Immunosuppression
* Active or systemic infection
* Collagen vascular disease
* Diabetes
* Venous stasis ulcers
* Participant undergoing active cancer chemotherapy
* Chronic steroid use
* Decision impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-07; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Wound healing over time | July 2008-October 2009

SECONDARY OUTCOMES:
Comparing three FDA cleared products for pain reduction and incidence of infection | July 2008-October 2009

CONTACTS AND LOCATIONS:
Overall Officials: Scott N Sheftel, MD, Principal Investigator — Sheftel Associates Dermatology, LLC
Locations (2):
- United States (2):
  - Sheftel Associates Dermatology, LLC, Oro Valley, Arizona
  - Sheftel Associates Dermatology, LLC, Tucson, Arizona